CLINICAL TRIAL: NCT01503931
Title: Endophenotyping With fMRI: Genetic Modulation and Treatment Response
Brief Title: Endophenotyping With Functional Magnetic Resonance Imaging (fMRI)
Acronym: NGFN PLUS TP13
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Central Institute of Mental Health, Mannheim (Other); University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Andreas Heinz, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: 01GS08159
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence, functional magnetic resonance imaging, genetics, endophenotypes, dopamine,; glutamate
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood (EDTA)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Alcohol-dependent patients: * men and women, aged 18 to 75
  * legally effective, written informed consent for participation within the study
  * right handedness
  * no other psychiatric disorder according to ICD 10
  * no psychotropic substances within the last 7 days
- Healthy control subjects: * men and women, aged 18 to 75
  * legally effective, written informed consent for participation within the study
  * right handedness
  * no psychiatric disorder according to ICD 10
  * no psychotropic substances within the last 7 days

SUMMARY:
The mesolimbic dopaminergic reward system is a key structure underlying addictive behaviour in alcohol addiction and is under control of prefrontal glutamatergic neurotransmission. The aim of the present multicenter-study in Berlin, Bonn and Mannheim is to use functional magnetic resonance imaging (fMRI) in alcohol addiction for endophenotyping in order to study the relevance of genetic variation, in particular in dopaminergic and glutamatergic genes, for addiction. The investigators will use a temporal discounting and a cue reactivity paradigm in alcoholics and healthy controls in order to 1) test the impact of genetic variation on activation of the mesolimbic system in these populations and to 2) to test their predictive effects for treatment outcome in alcoholics. The subproject will thus bridge animal research on genetically determined cue reactivity and human studies in alcoholics. Furthermore, the investigators will link these results to the measurement of glutamate and glutamine with magnetic resonance spectroscopy (MRS) in subproject SP14.

DETAILED DESCRIPTION:
Alcohol addiction is one of the most common neuropsychiatric diseases in today's society. Chronic misuse of alcohol not only causes significant physical and psychological damage in afflicted individuals, it also represents a serious social and economic problem. Despite the availability of a range of psychological and medical therapies, the risk of relapse for dependent individuals remains high even after years of abstinence. New, more effective therapies are urgently needed. Approximately 50% of the predisposition to develop an alcohol addiction is genetically inherited. In order to create improved treatment approaches and novel diagnostic tools, an enhanced knowledge of the genetic basis and biology of alcohol addiction is a prerequisite.

The aim of this multi-centre study is to investigate how and which genetic variations increase the risk for developing an alcohol-addiction. To achieve this, scientists in Berlin, Bonn and Mannheim will examine specific brain mechanisms that play important roles in alcohol dependence. Functional Magnetic Resonance Imaging (fMRI), a technique that makes it possible to observe the brain 'at work', will be used to reveal brain mechanisms affected by alcohol addiction such as the processing of reward and punishment, behaviour control and memory. It will then be investigated which genes or gene-gene interactions underlie these neuronal mechanisms. This powerful approach has the potential to uncover 'addiction-pathways' through which genes affect personality, drinking behaviours and success in staying abstinent via their influences on neuronal mechanisms.

A special emphasis of this project lies upon the so-called 'reward system', which processes naturally rewarding stimuli (e.g. food, sex) and which, in alcohol-dependent individuals, changes perceptions and behaviours in such a way that they become progressively more focused on alcohol. Two major neurotransmitters are involved in the workings of the reward system: 'dopamine' and more indirectly 'glutamate'. The project will investigate how dopaminergic and glutamatergic genes influence the neural mechanisms of reward processing, other neural mechanisms, personality, drinking behaviours and therapy success. In the long run, this knowledge might lead to more effective therapies such as the development of new medications.

This large-scale study will be conducted with several hundreds of alcohol-dependent patients and non-dependent individuals over a period of five years.

ELIGIBILITY:
Inclusion Criteria:

Healthy Controls

* men and women, aged 18 to 75
* legally effective, written informed consent for participation within the study
* right handedness
* no psychiatric disorder according to ICD 10
* no psychotropic substances within the last 7 days Alcohol-dependent patients
* men and women, aged 18 to 75
* legally effective, written informed consent for participation within the study
* right handedness
* no other psychiatric disorder according to ICD 10
* no psychotropic substances within the last 7 days

Exclusion Criteria:

* physical disorders, which might interfere with the planned examination (e.g. cerebral or organic disorder)
* MR-contraindication (z.B. pace maker, metalic or electronic implants, metal splinters, operation clips)
* anamnestic manifest psychiatric axis I disorder and/or axis II according to ICD-10 except alcohol dependence for patients
* medication or drug dependence
* medication or drug abuse (randomized urin testing)
* insufficient knowledge of German language
* claustrophobia
* for women: pregnancy (exclusion via pregnancy test)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2008-06; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
blood oxygenation level dependent (BOLD) response | first assessment timepoint (alc.dep. patients: up to 21 days after detoxification)
  investigation of neuronal activation of the mesolimbic system in alcohol-dependent patients and healthy controls using 3 tesla magnetic resonance imaging
Genetic endophenotypes | second assessment timepoint: 3 days after first assessment time point
  study the relevance of genetic variation, in particular in dopaminergic and glutamatergic genes, for addiction

SECONDARY OUTCOMES:
Treatment response | 6 month follow up period beginning after second assessment timepoint
  test the predictive effects of endophenotypes (genetic and imaging factors) for treatment outcome (relapse vs. abstinence) in alcohol-dependent patients

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Heinz, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Dept. of Psychiatry and Psychotherapy, Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Jorde A, Bach P, Witt SH, Becker K, Reinhard I, Vollstadt-Klein S, Kirsch M, Hermann D, Charlet K, Beck A, Wimmer L, Frank J, Treutlein J, Spanagel R, Mann K, Walter H, Heinz A, Rietschel M, Kiefer F. Genetic variation in the atrial natriuretic peptide transcription factor GATA4 modulates amygdala responsiveness in alcohol dependence. Biol Psychiatry. 2014 May 15;75(10):790-7. doi: 10.1016/j.biopsych.2013.10.020. Epub 2013 Nov 4. PMID 24314346
- See also: Homepage of the project (NGFN PLUS TP 13) — http://www.ngfn.de/en/tp13_endoph__notypisierung_alkoholabh__ngiger_patienten_mit_fmrt__genetische_modulation_und_behandlungsresponse.html